CLINICAL TRIAL: NCT03730246
Title: Postoperative Pain 0-24 hr After Cesarean Sectio
Brief Title: Pain After Cesarean Sectio.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Johan C Ræder, Professor, Oslo University Hospital
Other Study IDs: Sectio.Pain.Jenny
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Pain; Analgesic Medication
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cesarean sectio — consecutive parturients due for cesarean sectio

SUMMARY:
To study the strength of postoperative pain 0-24 hrs after elective cesarean sectio in spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* cesearean sectio

Exclusion Criteria:

* none

Max Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: all patients due for cesarean sectio are eligible
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
postoperative pain strenght | 0-24 hrs
  NRS pain

SECONDARY OUTCOMES:
rescue drug needed | 0-24 hrs
  dose of rescue opioid drug

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Anesthesiology, Oslo University Hospital, Ullevaal, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No